CLINICAL TRIAL: NCT03584867
Title: Scheduled CPR Refresher Training Role in Retaining Psychomotor Skills
Brief Title: CPR Refresher Role in Retaining Psychomotor Skills
Acronym: RefCPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SQU-EC/023/18
Record Dates: First submitted 2018-03-07; First posted 2018-07-12 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Arrest
Keywords: Basic life support; CPR skills; Training; High quality CPR
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Randomized controlled study. Experimental group would receive a refresher training at six months wherease the control receive not training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study Group (Experimental): refresher CPR
  Interventions: Other: refresher training at six months
- control (No Intervention): NO refresher

INTERVENTIONS:
Other: refresher training at six months — a 5 cycles of 30:2 compression to ventilation ratio will be offered to experimental group at six months from BLS certification.
  Arms: study Group

SUMMARY:
The study aims to measure the effectiveness of refresher training after six months of baseline training on retention of CPR skills. Literature review and guidelines showed that there is significant decay in CPR skills after basic life support certification. This retention might be preserved as short as three months after basic life support certification. Frequent retraining within the standard two years of recertification was recommended. Recommendation did not specify the ideal timing and method for CPR refresher training. In this study, we are looking for a feasible, practical, easily applicable method for health care institute in order to maintain the required CPR skills. This study will be a randomized control trial in which the study group will be tested for their CPR skills at six and twelve months after CPR training before the start of the study and after six months assessment. The control group will be tested after twelve months from the initial training at the start of the research and with no CPR refresher in between. The outcome of the study will assess the effectiveness of a BLS refresher training at six months on retention of quality of CPR skills.

DETAILED DESCRIPTION:
This is a prospective study that will enrol nurses, doctors and respiratory therapists of the Sultan Taboos university hospital,emergency departments from February 2018 until February 2019. All participants will be verbally consented before enrolment. Participants can withdraw from the study at any stage. All subjects will be assessed initially for their baseline skills of CPR. Assessment will be through measuring the baseline performance of the subjects. This will be two minutes of CPR in which chest compression rate, depth, chest recoil, interruption and ventilation will be assessed. CPR meter device will be used in each CPR assessment throughout the study. After that, all participants will receive CPR training which includes 15minutes standard CPR video followed by five minutes instructor- led teaching in manikins. Individual CPR performance will be assessed for each subject and data will be collected using a standardized data collection sheet. Next, groups will be randomized into two different groups using stratified sampling method to account for the years of experience. Participants will be divided into groups based on experience; 0-5, 5-10, 10-15, 15-20 and more than 20 years. Research randomizer (https://www.randomizer.org) program will be used for this purpose. Then, subjects will be randomized into study(group1) and control(group2) group. Both groups will be called after 6 months. Pre-assessment test will be conducted, which is similar to the baseline assessment test, for both groups using the same standardized data collection sheet. Then, study group will receive refresher training of CPR while the control group will be released with no training. Six months later, both groups will be called and CPR skills will be assessed again.

CPR performance will be monitor and assessed by using Little Anne manikin which has quality CPR (QCPR) monitoring through smart devises. This will provide data for each performer including chest compression rate and depth, chest recoil and adequate ventilation. Data of each subject will be stored in the devise and then will be transferred to software for storage and analysis.

ELIGIBILITY:
Inclusion Criteria:

* All sultan Taboos university hospital staff in emergency department( nurses, doctors and respiratory therapists) who received basic life support training
* Age more than 18 years old

Exclusion Criteria:

* Medical illnesses that interfere with chest compression (back pain, wrist pain, knee pain)
* Pregnancy
* Providers who are scheduled for refresher training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Chest compression | 12 months
  Chest compression rate ( number of compression per minute) Descriptive statistics will be presented as a mean ± standard deviation by using student t-test

SECONDARY OUTCOMES:
Ventilation rate | 12 months
  adequate or not adequate
time of interruption | 12 months
  measured in seconds
depth of compression | 12 months
  measured in millimetres

CONTACTS AND LOCATIONS:
Overall Officials: Mahmood AlJufaili, M.D., Principal Investigator — Sultan Qaboos University
Locations (2):
- Oman (2):
  - Sultan Qaboos University, Muscat
  - Sultan Qaboos university hospital, Muscat

IPD SHARING:
Plan to Share IPD: No
Confidentiality issue

REFERENCES:
- [Result] Jensen ML, Lippert F, Hesselfeldt R, Rasmussen MB, Mogensen SS, Jensen MK, Frost T, Ringsted C. The significance of clinical experience on learning outcome from resuscitation training-a randomised controlled study. Resuscitation. 2009 Feb;80(2):238-43. doi: 10.1016/j.resuscitation.2008.10.026. Epub 2008 Dec 5. PMID 19058890
- [Result] Niles D, Sutton RM, Donoghue A, Kalsi MS, Roberts K, Boyle L, Nishisaki A, Arbogast KB, Helfaer M, Nadkarni V. "Rolling Refreshers": a novel approach to maintain CPR psychomotor skill competence. Resuscitation. 2009 Aug;80(8):909-12. doi: 10.1016/j.resuscitation.2009.04.021. Epub 2009 May 20. PMID 19467759
- [Result] Yang CW, Yen ZS, McGowan JE, Chen HC, Chiang WC, Mancini ME, Soar J, Lai MS, Ma MH. A systematic review of retention of adult advanced life support knowledge and skills in healthcare providers. Resuscitation. 2012 Sep;83(9):1055-60. doi: 10.1016/j.resuscitation.2012.02.027. Epub 2012 Mar 3. PMID 22391016
- [Result] Nishiyama C, Iwami T, Murakami Y, Kitamura T, Okamoto Y, Marukawa S, Sakamoto T, Kawamura T. Effectiveness of simplified 15-min refresher BLS training program: a randomized controlled trial. Resuscitation. 2015 May;90:56-60. doi: 10.1016/j.resuscitation.2015.02.015. Epub 2015 Feb 24. PMID 25724354
- [Result] Oermann MH, Kardong-Edgren SE, Odom-Maryon T. Effects of monthly practice on nursing students' CPR psychomotor skill performance. Resuscitation. 2011 Apr;82(4):447-53. doi: 10.1016/j.resuscitation.2010.11.022. Epub 2011 Jan 11. PMID 21227563
- [Result] Kardong-Edgren SE, Oermann MH, Odom-Maryon T, Ha Y. Comparison of two instructional modalities for nursing student CPR skill acquisition. Resuscitation. 2010 Aug;81(8):1019-24. doi: 10.1016/j.resuscitation.2010.04.022. Epub 2010 Jun 2. PMID 20566391
- [Result] Niles DE, Nishisaki A, Sutton RM, Elci OU, Meaney PA, O'Connor KA, Leffelman J, Kramer-Johansen J, Berg RA, Nadkarni V. Improved Retention of Chest Compression Psychomotor Skills With Brief "Rolling Refresher" Training. Simul Healthc. 2017 Aug;12(4):213-219. doi: 10.1097/SIH.0000000000000228. PMID 28368963
- [Result] Soar J, Monsieurs KG, Ballance JH, Barelli A, Biarent D, Greif R, Handley AJ, Lockey AS, Richmond S, Ringsted C, Wyllie JP, Nolan JP, Perkins GD. European Resuscitation Council Guidelines for Resuscitation 2010 Section 9. Principles of education in resuscitation. Resuscitation. 2010 Oct;81(10):1434-44. doi: 10.1016/j.resuscitation.2010.08.014. No abstract available. PMID 20956044
- [Result] Sutton RM, Nadkarni V, Abella BS. "Putting it all together" to improve resuscitation quality. Emerg Med Clin North Am. 2012 Feb;30(1):105-22. doi: 10.1016/j.emc.2011.09.001. Epub 2011 Oct 15. PMID 22107978
- [Result] Meaney PA, Bobrow BJ, Mancini ME, Christenson J, de Caen AR, Bhanji F, Abella BS, Kleinman ME, Edelson DP, Berg RA, Aufderheide TP, Menon V, Leary M; CPR Quality Summit Investigators, the American Heart Association Emergency Cardiovascular Care Committee, and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. Cardiopulmonary resuscitation quality: [corrected] improving cardiac resuscitation outcomes both inside and outside the hospital: a consensus statement from the American Heart Association. Circulation. 2013 Jul 23;128(4):417-35. doi: 10.1161/CIR.0b013e31829d8654. Epub 2013 Jun 25. PMID 23801105
- [Result] Bhanji F, Donoghue AJ, Wolff MS, Flores GE, Halamek LP, Berman JM, Sinz EH, Cheng A. Part 14: Education: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S561-73. doi: 10.1161/CIR.0000000000000268. No abstract available. PMID 26473002